CLINICAL TRIAL: NCT06264908
Title: Hand OsteoArthritis Self-management and Integrated Scheme (OASIS-H) to Improve Outcomes in Patients With Hand Osteoarthritis
Brief Title: An Integrated Self Management Programme to Improve Outcomes in Patients With Hand Osteoarthritis
Acronym: OASIS-H
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Iris Tang Yan Ki (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Sponsor-Investigator, Dr Iris Tang Yan Ki, Clinical Assistant Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20240125-010-000
Record Dates: First submitted 2024-01-31; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hand Osteoarthritis
Keywords: hand osteoarthritis; self-management programme

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into early intervention and routine clinical care (control) group. Patients in control group will crossover to receive the intervention at week 26.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early intervention arm (Experimental): 8 weeks integrated self-management programme delivered by occupational therapists and rheumatology nurse
  Interventions: Behavioral: Integrated self-management programme
- Routine Clinical care (Control) (No Intervention): Patients will receive routine clinical care for hand osteoarthritis for 26 weeks, then cross-over to the integrated programme after 26 weeks.

INTERVENTIONS:
Behavioral: Integrated self-management programme — 8 weeks integrated management programme with three educational sessions. Group therapy sessions (6-8 participants per group) delivered by occupational therapists and rheumatology nurses.
  1. Disease pathology and Pain management
  2. Joint protection and stretching exercise
  3. Psychosocial education
  4. Aids prescription Each session will consist of education session, exercise session and group sharing sessions.
  Arms: Early intervention arm

SUMMARY:
The goal of this trial is to evaluate the efficacy of an integrated self-management programme in improving clinical outcomes in patients with hand osteoarthritis (OA).

This is an open-labelled, randomized controlled trial with an objective to determine the efficacy of an integrated self-management programme versus routine clinical care for participants with symptomatic hand OA.

Participants will be randomized into early intervention group and routine clinical care groups in a 1:1 ratio. Patients who randomized into early intervention group will receive 8 week integrated self-management programme delivered by occupational therapists and rheumatology nurse on hand OA management. Patients who randomized into routine clinical care group will receive usual clinical care for OA for 26 weeks and then receive an identical 8 weeks integrated self-management programme. The primary outcome is the improvement in pain at 26 weeks between the two groups.

DETAILED DESCRIPTION:
Background: Osteoarthritis (OA) of the hand is a common and potentially disabling condition with increasing prevalence in Hong Kong due to an aging population. The direct and indirect economic burden due to OA are substantial and this calls for an unmet need for more effective management for hand OA. Hand OsteoArthritis Self-management and Integrated Scheme (OASIS-H) is a self-management programme integrated with occupational therapy and rheumatology nurse education with an aim to improve outcomes in patients with hand osteoarthritis.

Objective: This is an open-labelled, randomized controlled trial to determine the efficacy of an integrated self-management programme versus routine clinical care for participants with symptomatic hand OA.

Hypothesis: The integrated programme will be more efficacious than routine clinical care in reducing pain and improving function in symptomatic OA hand in 6 months.

Methods: Consecutive patients who fulfilled the American College of Rheumatology Classification Criteria for hand OA with a pain score of ≥40 out of 100mm on visual analogue scale (VAS) will be included. Patient with secondary OA hand, unable to sign consent and with the use of systemic corticosteroid within 6 months will be included. Participants will be randomized in a 1:1 ratio into early intervention and routine clinical care groups. In the early intervention group, patients will participate in an eight-week integrated hand OA management programme within 1 month from randomization. The programme will consist of three self-management education sessions conducted by the occupational therapists and rheumatology nurses on pain management strategy, joint protection, group sharing and exercise, one telemedicine session, aids prescription and splintage fabrication. For patients randomized into the routine clinical care group, they will continue to receive routine medical care from the rheumatology clinic. At 6 months after randomization, patients in the routine clinical care group will crossover and receive an identical 8-week integrated hand OA management programme as the early intervention group. The primary endpoint is the change in finger pain in pain VAS at 6 months from baseline. Secondary endpoints include change in function measured by the functional index for functional index for hand OA, Short form health survey and health assessment questionnaire disability index, change in hand grip strength and dexterity at 6 months and 12 months. The primary endpoint will be analyzed by linear mixed models and the differences in pain over time between the two groups will be compared using linear regression model.

ELIGIBILITY:
Inclusion Criteria:

* Fulfil the American College of Rheumatology hand osteoarthritis classification criteria
* Symptomatic hand osteoarthritis with a pain visual analogue score (VAS) equal to or more than 40/100mm within 2 weeks of study entry

Exclusion Criteria:

* Secondary hand osteoarthritis from inflammatory arthritis including rheumatoid arthritis, spondyloarthropathy, psoriatic arthritis, gouty arthropathy or connective tissue diseases;
* Receive systemic corticosteroids (other than topical or inhalational) within 6 months of study entry
* Inability to sign informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Change in Pain visual analogue scale (VAS) | 26 weeks
  Pain VAS reflects the severity of pain in a score of 0-100. A lower score indicates less pain.

SECONDARY OUTCOMES:
Change in pain Visual Analogue Scale (VAS) | 12weeks, 52 weeks
  Pain VAS reflects the severity of pain in a score of 0-100. A lower score indicates less pain.
Change in Functional index hand osteoarthritis (FIHOA) | 12 weeks, 26 weeks, 52 weeks
  FIHOA reflects hand function with a score of 0 to 30. A lower score indicates better hand function
Change in Quick Disabilities of the Arm, Shoulder, and Hand (DASH) score | 12 weeks, 26 weeks, 52 weeks
  QuickDASH is a self-reported 11-itemed questionnaire in which the response options are presented as 5-point Likert scales. At least 10 of the 11 items must be completed for a score to be calculated and the scores range from 0 (no disability) to 100 (most severe disability)
Change in Australian/Canadian Hand Osteoarthritis Index (AUSCAN) 3.1 | 12 weeks, 26 weeks, 52 weeks
  AUSCAN 3.1 hand osteoarthritis index is a self-administered questionnaire that assesses the three dimensions of pain, disability and joint stiffness in hand osteoarthritis using a battery of 15 questions. The score is expressed in 3 subscores: AUSCAN pain score (0 (least painful)-100 (most painful), the AUSCAN stiffness score (0: least stiffness-100: most stiffness), the AUSCAN function score (0: least function impairment-100: most severe function impairment)
Change in Short-form 36 items health survey | 26 weeks, 52 weeks
  Short-form 36 items health survey measures 8 domains of health related quality of life. The score is expressed in 0 - 100. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change in hand grip strength | 26 weeks, 52 weeks
  Hand grip strength measured by dynamometer
Change in hand dexterity measurement | 26 weeks, 52 weeks
  Hand dexterity measurement
Radiographic changes | 52 weeks
  Measured by hand plain radiographs

OTHER OUTCOMES:
Adverse events | up to 52 weeks
  Adverse events
Use of rescue pain medication | up to 52 weeks
  Use of rescue pain medication e.g. NSAIDS / steroids

IPD SHARING:
Plan to Share IPD: No